CLINICAL TRIAL: NCT05561335
Title: Comparison of a Novel Algorithm to a Standard Microphone Configuration for Hearing Preference
Brief Title: Preference Comparisons for Algorithms to Hear Speech
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sonova AG (Industry)
Collaborators: Western University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5251
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearing Aid use for listening to speech in a common difficult situation (Experimental): The hearing aids will be worn in two different programs, each with a different microphone configuration. The participants will listen to speech while wearing the hearing aids and alternate programs to form their opinions about these programs; they will only know that they are rating different settings, not what the settings are. They will then rate their listening experiences via rating scales to determine their preferences.
  Interventions: Device: hearing aid -novel program; Device: hearing aid - standard program

INTERVENTIONS:
Device: hearing aid -novel program — novel microphone configuration
Device: hearing aid - standard program — standard microphone configuration

SUMMARY:
Twenty people with hearing impairment will be tested and fitted binaurally with hearing aids. During a real-world listening situation, each participant will be asked to compare one program with a novel algorithm to one with a standard microphone configuration. They will provide ratings on a range of outcome measures including overall preference and awareness of background noise. Overall and specific preferences for the different programs/algorithms will be determined by their subjective responses to determine if there is a significant difference between the two programs.

DETAILED DESCRIPTION:
People with hearing loss/impairment often have difficulty not only hearing certain sounds (e.g., environmental and speech sounds) but also listening in certain situations such as those where noise competes with speech. This is a common situation in people's real life conversations and one which different hearing instrument algorithms could facilitate.

This study will investigate the listening preferences of people with hearing impairment while wearing hearing aids. They will listen to speech in a situation which is commonly reported as difficult for people who wear hearing aids. Participants will wear one set of hearing aids set to their hearing loss with two programs providing these different algorithms. By having the participants toggle (with a remote control) back and forth between algorithms designed for these real-life difficult listening situations, they can rate their preferences and listening experiences.

Of particular interest, in addition to overall preference, are ratings of the background noise, listening effort and annoyance of artefacts.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling all of the following inclusion criteria are eligible for the investigation:

* Including adults with sensorineural mild to moderate-severe hearing loss
* hearing aid experience (greater than 6 months)
* who are able to complete the task in English.
* Language: Can speak and understand English Fluently

Hearing loss within the fitting ranges of the investigational products.

* Healthy outer ear.
* Ability to understand instructions.
* Ability to describe listening experiences.
* Ability to fill out questionnaires.
* Informed consent as documented by signature.

Exclusion Criteria:

- The presence of any one of the following exclusion criteria will lead to the exclusion of the subject:

* Contraindications to the MD in this study (e.g. known hypersensitivity or allergy to the investigational product).
* Limited mobility and not able to attend to appointments or not able to go in a car.
* Reported symptoms of vertigo and dizziness by subject.
* Severe Tinnitus

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall preference for a specific microphone setting/configuration | 20 minutes
  Rating of preference on a scale from 0-100, with descriptors ('very low' to 'very high')

SECONDARY OUTCOMES:
Rating of awareness of background noise | 20 minutes
  Scale from 0-100 with descriptors ('not at all' to 'extremely aware')
Rating of Listening effort | 20 minutes
  Scale from 1 - 7 with descriptors ('not at all' to 'very')
Rating of annoyance of artefacts | 20 minutes
  Rating on a scale from 0-100 with descriptors ('not at all' to 'extremely annoying')

CONTACTS AND LOCATIONS:
Overall Officials: Susan Scollie, PhD, Principal Investigator — Western University (aka The University of Western Ontario)
Locations (1):
- Western University, London, Ontario, Canada